CLINICAL TRIAL: NCT00749255
Title: R2 Case Collection
Brief Title: Collect Breast Cancer Patients' Digital Mammography Images With Corresponding Reports for the Development of Software
Status: Terminated | Type: Observational
Why Stopped: not enough personnel to conduct study at site
Sponsor: WellSpan Health (Other)
Responsible Party: Misty Hicks, RTRM, Women's Imaging
Other Study IDs: 0708052
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Digital archiver software
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FFDM: a sum of at least 200 cancer cases, mammographically visible, on at least one image view (including masses and calcifications)

SUMMARY:
The purpose of this case collection effort is software design by R2 Technologies, Inc., The information received from Women's Imaging will be provided to the Case Collection, Data Management and Algorithm/software design and development teams who are responsible for the receipt of patient data and management of such data; and creation, testing and validation of R2 Technologies, Inc., for Computer Aided Detection (CAD) and new digital image archiving software design.

DETAILED DESCRIPTION:
The information is necessary for Sponsor development efforts and will be utilized as a viewing tool with supporting written documentation of the findings on each image itself. The information will be used to develop algorithms that will foster development of CAD software. The information in each image and/or accompanying written clinical case documentation will not be analyzed in any way for clinical events

ELIGIBILITY:
Inclusion Criteria:

* subjects with known breast cancer ages 18 and over
* case images originating from Women's imaging or one of the affiliated screening centers. Raw images must be available for each image
* source documents or mammographic interpretation must be available

Exclusion Criteria:

* 17 or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Known breast cancer patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-05; Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misty Hicks, RTRM, Principal Investigator — Women's Imaging @ WellSpan Health
Locations (1):
- Women's Imaging @ WellSpan Health, York, Pennsylvania, United States